CLINICAL TRIAL: NCT07298460
Title: Transcutaneous Spinal Cord Stimulation to Improve Postural Stability After Surgery for Degenerative Cervical Myelopathy
Brief Title: Stimulation-based Therapy to Improve Balance in DCM
Acronym: STIM-DCM
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other); Advancing a Healthier Wisconsin Endowment (Unknown); Froedtert Hospital (Other)
Responsible Party: Principal Investigator, Aditya Vedantam, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Cervical Myelopathy
Keywords: degenerative cervical myelopathy; spinal cord stimulation; balance; therapy; rehabilitation; postural instability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Thoracic tSCS + balance training (Active Comparator): This intervention combines noninvasive thoracic transcutaneous spinal cord stimulation (tSCS) with a structured balance training program specifically for adults with degenerative cervical myelopathy (DCM) who have undergone surgical decompression but continue to experience impaired balance.
  Interventions: Device: Transcutaneous spinal cord stimulation; Other: Balance and Gait Training
- Combined cervical and thoracic tSCS + balance training (Active Comparator): This intervention combines noninvasive combined cervical and thoracic transcutaneous spinal cord stimulation (tSCS) with a structured balance training program specifically for adults with degenerative cervical myelopathy (DCM) who have undergone surgical decompression but continue to experience impaired balance.
  Interventions: Device: Transcutaneous spinal cord stimulation; Other: Balance and Gait Training
- Sham tSCS + balance training (Sham Comparator): This intervention combines sham transcutaneous spinal cord stimulation (tSCS) with a structured balance training program specifically for adults with degenerative cervical myelopathy (DCM) who have undergone surgical decompression but continue to experience impaired balance.
  Interventions: Other: Balance and Gait Training

INTERVENTIONS:
Device: Transcutaneous spinal cord stimulation — This intervention combines noninvasive transcutaneous spinal cord stimulation (tSCS) with a structured balance training program specifically for adults with degenerative cervical myelopathy (DCM) who have undergone surgical decompression but continue to experience impaired balance. Unlike standard physical therapy or other neuromodulation approaches, this protocol uses targeted stimulation sites and parameters-thoracic-only or combined cervico-thoracic stimulation-delivered concurrently with task-specific balance and gait training to enhance neuromotor recovery. The stimulation is applied using a Chattanooga Vectra device at tolerable intensity, integrated into 12 sessions over 4 weeks. This design uniquely addresses persistent postural instability in post-surgical DCM.
  Arms: Combined cervical and thoracic tSCS + balance training; Thoracic tSCS + balance training
Other: Balance and Gait Training — Structured balance and gait training will be performed for the participant.

SUMMARY:
The goal of this clinical trial is to determine if a treatment called transcutaneous spinal cord stimulation (tSCS), when combined with balance training, can help improve balance in adults who have had surgery for degenerative cervical myelopathy (DCM). DCM is a condition that affects the spinal cord in the neck and often causes problems with walking and balance, even after surgery.

This study will also look at how tSCS affects the nervous system and whether it is safe and practical to use in this group of patients. The results will help researchers plan a larger study in the future.

Main Questions:

* Does tSCS combined with balance training improve balance more than balance training alone?
* Does stimulation at both the neck and mid-back work better than stimulation at the mid-back only?
* What changes in nerve and muscle activity occur with tSCS?

What will happen in this study:

* Participants will be randomly assigned to one of three groups:

  1. tSCS applied to the mid-back (thoracic area) plus balance training
  2. tSCS applied to both the neck and mid-back (combined stimulation) plus balance training
  3. Sham stimulation (electrodes placed but no stimulation) plus balance training
* All participants will complete 12 sessions over 4 weeks (3 sessions per week).
* Each session will include 30 minutes of balance training and 30 minutes of walking exercises.
* Participants will receive stimulation or sham treatment during these sessions.
* Balance and walking tests will be done before and after the program.
* Nerve and muscle activity will also be measured at the same time points.

This pilot study will help determine if tSCS is effective and safe, and will provide information needed to design a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* DCM participants who have undergone surgery for DCM more than 12 months prior and report persistent impaired imbalance

Exclusion Criteria:

* uncontrolled cardiopulmonary disease, legal blindness, unstable medical condition that can interfere with the study, breakdown in skin area that will come into contact with electrodes, active implanted medical device, pregnancy, and seizures
* concurrent occupational or physical therapy during study participation for any condition
* history of inability to tolerate MEP/SSEP for any reason, or complete paralysis of the legs (lower limb mJOA=0)
* cognitive impairment and unable to give consent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | From enrollment to the end of the intervention at 4 weeks
  The Berg Balance Scale is a validated clinical measure of static and dynamic balance.
Motor evoked potential (MEP) amplitude in the quadriceps of either leg | From enrollment to the end of the intervention at 4 weeks
  Motor evoked potential (MEP) amplitude recorded from the quadriceps to assess changes in corticospinal excitability when comparing combined cervico-thoracic tSCS versus thoracic-only tSCS.

SECONDARY OUTCOMES:
Center of pressure (CoP) path length and mean velocity during the modified Clinical Test of Sensory Integration for Balance (mCTSIB) with eyes closed on firm and foam surfaces | From enrollment to the end of the intervention at 4 weeks
  Total displacement of the center of pressure during quiet standing with eyes closed on firm and foam surfaces, reflecting postural sway magnitude.
Sensory Organization Test (SOT) - Somatosensory and Vestibular Score | From enrollment to the end of the intervention at 4 weeks
  Quantifies reliance on somatosensory and vestibular input for balance under altered sensory conditions.
Single-Leg Stance Time | From enrollment to the end of the intervention at 4 weeks
  Duration of stable single-leg standing, assessing unilateral static balance capacity.
Functional Gait Assessment (FGA) | From enrollment to the end of the intervention at 4 weeks
  Performance-based measure of dynamic balance during complex walking tasks.
6-Meter Walk Test Gait Speed | From enrollment to the end of the intervention at 4 weeks
  Average walking speed over a short distance, reflecting functional mobility and gait efficiency.
Timed Up and Go (TUG) | From enrollment to the end of the intervention at 4 weeks
  Time required to stand, walk, turn, and sit, capturing functional mobility and fall risk.
Responder Status (MCID Achievement) | From enrollment to the end of the intervention at 4 weeks
  Proportion of participants achieving a minimum clinically important improvement in predefined outcomes.
Modified Japanese Orthopaedic Association (mJOA) Score | From enrollment to the end of the intervention at 4 weeks
  Clinician-rated measure of neurological function in cervical myelopathy.
Neck Disability Index (NDI) | From enrollment to the end of the intervention at 4 weeks
  Patient-reported measure of neck-related functional disability.
Numeric Rating Scale (NRS) for Pain | From enrollment to the end of the intervention at 4 weeks
  Patient-reported pain intensity for neck, arm, leg, and device-related pain on a 0-10 scale.
SF-36 Physical Component Score (PCS) | From enrollment to the end of the intervention at 4 weeks
  Generic health-related quality-of-life measure focused on physical functioning.
Clinician Global Impression of Change (CGIC) | From enrollment to the end of the intervention at 4 weeks
  Clinician-rated assessment of overall change in patient condition.
Patient Global Impression of Change (PGIC) | From enrollment to the end of the intervention at 4 weeks
  Patient-reported perception of overall improvement or worsening.
Fall Frequency | From enrollment to the end of the intervention at 4 weeks
  Number of self-reported falls recorded prospectively in a fall diary.
Adverse Events (AEs) and Serious Adverse Events (SAEs) | From enrollment to the end of the intervention at 4 weeks
  Incidence and severity of treatment-emergent adverse and serious adverse events.
Lower-Extremity Somatosensory Evoked Potential (SSEP) Latencies | From enrollment to the end of the intervention at 4 weeks
  Cortical response latencies following peripheral stimulation, reflecting integrity and conduction efficiency of ascending somatosensory pathways.
Motor Evoked Potentials (MEPs) - Tibialis Anterior and Abductor Pollicis Brevis | From enrollment to the end of the intervention at 4 weeks
  Evoked motor responses assessing corticospinal tract excitability and conduction to the lower extremities.
Surface EMG Amplitude - Tibialis Anterior and Quadriceps | From enrollment to the end of the intervention at 4 weeks
  Magnitude of muscle activation during stimulation, indexing neuromuscular recruitment of ankle dorsiflexors and knee extensors.

CONTACTS AND LOCATIONS:
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study will not be shared publicly. De-identified data may be made available upon reasonable request to the corresponding investigator, subject to approval by the institutional review board and execution of a data use agreement.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data will be available after publication of the primary results and for up a particular duration thereafter. This time period will be determine by the IRB and data use agreement.
Access Criteria: De-identified individual participant data and supporting documentation (including the study protocol and statistical analysis plan) will be made available to qualified researchers upon reasonable request. Requests must include a methodologically sound research proposal and will be reviewed by the study investigators. Access will be granted following institutional review board approval, as applicable, and execution of a data use agreement. Data will be provided through a secure data-sharing mechanism.
URL: https://clinicaltrials.gov